CLINICAL TRIAL: NCT05074004
Title: The Effect of Psychoeducation Given In Psychiatry Day Hospital on The Self-Sufficiency and Well-Being of The Patients
Brief Title: The Effect of Psychoeducation Given In Psychiatry Day Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İlkay KESER, Assist. Prof. Dr, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0707
Record Dates: First submitted 2021-09-08; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Chronic Mental Disorder; Psychoeducation
Keywords: chronic mental disorder; self-sufficiency; well-being; psychoeducation; psychiatric nurse; Turkey

STUDY DESIGN:
Intervention Model Description: The research is a single-blind randomized controlled experimental study
Who Masked: Participant
Masking Description: In the envelope method, 15 envelopes with '1' symbolizing the intervention group and 15 envelopes with '2' symbolizing the control group were found in the box. All individuals pulled envelopes out of the box, and the envelope was not put in the box again. During the psychoeducation process, one patient from the experimental group did not want to continue the training, and one patient from the control group was hospitalized; two patients were excluded from the sample.The pretest evaluation was made in the first interview with the individuals included in the sample. Posttest evaluation was made at the end of the intervention to the individuals in the intervention group. No intervention was applied to the control group in this process. Posttest evaluation was made at the end of the 8th week following the pretest evaluation to the control group. After all evaluations were completed, a single-session informative training was given to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No intervention was applied to the control group in this process.
  * be receiving treatment in Clinic Day Hospital
  * Volunteering to participate in research
- Psychoeducation (Experimental): * be receiving treatment in Clinic Day Hospital
  * Volunteering to participate in research
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Psychoeducation — Psychoeducation sessions were conducted by two psychiatric nurses (İK, SS) who are experts in their fields and have psychoeducation and group leadership certificates. Each session was held once a week in 30-45 minutes sessions. The training was carried out interactively; approximately the first 5 minutes were spent on warm-up, the basic information of that day's session was given for 25 minutes, and the last 10 minutes were in the form of questions and answers. Two separate groups were formed according to the day hospital program of the patients, and the psychoeducation program was carried out in two separate groups to conduct psychoeducation effectively.
  Arms: Psychoeducation

SUMMARY:
Background: Psychoeducation is a process used in the realization of the principles of treatment and rehabilitation of mental illnesses and aims to help the patient and his/her family outside the hospital, to help the patient cope with the problems, experiencing, and to support them to live productive lives in society.

Aims: This study aims to determine the effect of psychoeducation, given in a psychiatry dayhospital, on patients' self-sufficiency and well-being.

Methods: The research is a single-blind randomized controlled experimental study. The sample of the study consisted of 28 schizophrenic patient(14experiment-14control), who agreed to participate in the study, followed in XXX University Psychiatry Day Hospital. In the study, an 8-week psychoeducation program was applied to the experimental group, and no intervention was made tothe control group. Socio-demographic data form, self-sufficiency scale, and well-being scale were used as data collection tools. The data obtained were analyzed using theSPSS-23 package program.

Results: After the eight-week psychoeducation program, the pretest and posttest scores of the evaluations obtained from the scales of both groups were compared. It was found that while there was no change in thescores of the control group, there was an increase in the well-being and self-efficacy scores of the experimental group. While the increase in well-being was statistically significant(p<0.05), the increase in self-sufficiency score wasnot statistically significant(p>0.05), but the numerical increase was considered tobe aclinically significant result.

DETAILED DESCRIPTION:
Mental illnesses cause deterioration in various areas of functionality such as personal care, family and social relations, communication, professional life, and leisure activities. Mental diseases that cause disability are common in society. Mental disorders such as depression, schizophrenia, bipolar disorder, obsessive-compulsive disorder are among the diseases that cause loss of ability.

Rehabilitation services are important in order to support the adaptation of chronic mental patients to treatment outside the institution and to maintain their role in society. Self-sufficiency is one of the important issues to be addressed in chronic diseases that cause disability. Self-sufficiency refers to the individual's perception of the ability to successfully perform a certain action, the ability to control events, and the potential to accomplish a certain job. Individuals with high self-sufficiency set more difficult goals for themselves and make more efforts to achieve their goals. Since self-esteem is affected in mental disorders, self-sufficiency may be low.

High self-sufficiency leads to an increase in well-being. It is very important for psychological well-being for the individual to realize their potential and live a happy life. In recent years, attention has been paid to the well-being of individuals with mental disorders. Research has found that high well-being reduces disease recurrences. Some studies have also found that well-being is associated with having a depressive mood and an inability to cope with stress.

In psychological or physical diseases, educational intervention programs structured to teach people about their diseases and their emotional responses to the disease, to develop coping skills, to adapt to the disease, and to cooperate with treatment are defined as psychoeducation . The purpose of interventions is to teach individuals how to cope with their problems by creating knowledge and behavior changes, to help the patient to understand their own situation, to improve self-care activities, to prevent complications, to increase well-being and quality of life.

Studies in the literature conducted with different groups reveal that psychoeducation increases psychological resilience and supports coping with stress and feeling good. There are studies examining the effectiveness of psychoeducation from different aspects given to psychiatric patients. However, there is no study examining the effect of psychoeducation to evaluate the well-being and self-sufficiency of individuals who are in the rehabilitation phase and receive psychiatric treatment. The findings to be obtained as a result of the study will make a significant contribution to the psychiatric care and monitoring provided in day hospitals and rehabilitation centers and will create a database for new studies.

Purpose and hypotheses of the study This study was carried out to determine the effect of psychoeducation given in psychiatric day hospitals on the self-sufficiency and well-being of patients.

H1 Psychoeducation given in the psychiatric day hospital increases the self-sufficiency of the patients.

H2 Psychoeducation given in the psychiatric day hospital improves the well-being of the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who were followed up in the psychiatry day hospital,
* accepted to participate in the study,
* signed the informed consent form, and were able to read

Exclusion Criteria:

* individuals indicating their desire to leave the study,
* the development of an attack requiring hospitalization,
* not attending education for more than two sessions.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Socio-demographic Data Form | pre-intervention
  The form prepared by the researchers using the literature contains questions about the health status and the sociodemographic characteristics of individuals diagnosed with psychiatric diseases, such as age, gender, marital status, and educational status.
General Self-Sufficiency Scale | pre-intervention
  The Turkish adaptation of the scale developed by Sherer et al. (1982) was carried out by Yıldırım & İlhan (2010). The scale with a 5-point Likert structure consists of 17 items. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16 and 17 are scored in reverse. The total score that can be obtained varies between 17 and 85, and the increase in the score indicates increased self-sufficiency belief. The scale was applied by Yıldırım & İlhan (2010) to 895 people aged 18 and over with at least five years of education. In the reliability study, the internal consistency coefficient was calculated as α = .80 for the whole scale and between .78 and .81 for each subscale.
Well-being Scale | pre-intervention
  The Turkish adaptation study of the Well-Being Scale developed by Diener et al. (2009) was carried out by Fidan and Usta (2013). The scale has a 7-point Likert structure. The highest score that can be obtained from the scale is 56, and the lowest score is 8. There are no reverse-scored items on the scale. High scores from the scale indicate that the relevant individual has a high level of well-being. The reliability study of the scale was conducted by Fidan and Usta (2013) on a total of 385 high school 4th-grade students, 166 (43%) female and 219 (57%) male. The Cronbach alpha internal consistency coefficient of the Well-Being Scale was reported as .83.

SECONDARY OUTCOMES:
General Self-Sufficiency Scale: | immediately after the interventio
  The Turkish adaptation of the scale developed by Sherer et al. (1982) was carried out by Yıldırım & İlhan (2010). The scale with a 5-point Likert structure consists of 17 items. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16 and 17 are scored in reverse. The total score that can be obtained varies between 17 and 85, and the increase in the score indicates increased self-sufficiency belief. The scale was applied by Yıldırım & İlhan (2010) to 895 people aged 18 and over with at least five years of education. In the reliability study, the internal consistency coefficient was calculated as α = .80 for the whole scale and between .78 and .81 for each subscale.
Well-being Scale: | immediately after the interventio
  The Turkish adaptation study of the Well-Being Scale developed by Diener et al. (2009) was carried out by Fidan and Usta (2013). The scale has a 7-point Likert structure. The highest score that can be obtained from the scale is 56, and the lowest score is 8. There are no reverse-scored items on the scale. High scores from the scale indicate that the relevant individual has a high level of well-being. The reliability study of the scale was conducted by Fidan and Usta (2013) on a total of 385 high school 4th-grade students, 166 (43%) female and 219 (57%) male. The Cronbach alpha internal consistency coefficient of the Well-Being Scale was reported as .83.

CONTACTS AND LOCATIONS:
Overall Officials: İlkay Keser, Study Director — Akdeniz Universty
Locations (1):
- Akdeniz Universty Faculty of Nursing, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
research can be viewed by all researchers
Supporting Information: Study Protocol
Time Frame: ten years
Access Criteria: in search for keywords

REFERENCES:
- [Result] Kizilirmak Tatu M, Demir S. Effect of Group Psychoeducation on Treatment Adherence, Quality of Life and Well-Being of Patients Diagnosed with Schizophrenia. Issues Ment Health Nurs. 2021 Mar;42(3):256-266. doi: 10.1080/01612840.2020.1793244. Epub 2020 Aug 12. PMID 32783665